CLINICAL TRIAL: NCT06546566
Title: Effects of Video Game-Based and Conventional Breathing Exercises on Pulmonary and Extrapulmonary Features in Children with Asthma: a Randomized Comparative Study
Brief Title: Video Game-Based and Conventional Breathing Exercises on Pulmonary and Extrapulmonary Features in Children with Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: auhucgun03
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Asthma in Children
Keywords: asthma; children; conventional breathing exercises; video game-based breathing exercise; pulmonary function; respiratory muscle strength; peripheral muscle strength; functional capacity; quality of life; asthma control
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Patients in the experimental group will receive video game-based breathing exercises training for 8 weeks, 5 days a week, 30 minutes a day. The exercise program will consist of 5 breathing games included in the BreathingLabs game kit and each game will be performed in 2 sets of 10 repetitions. In addition to video game-based breathing exercises, coughing techniques and relaxation techniques will be taught and physical activity recommendations will be given.
  Interventions: Other: Video Game-Based Breathing Exercises
- Control Group (Active Comparator): Patients in the control group will receive home-based conventional breathing exercises training for 8 weeks, 5 days a week, 30 minutes a day. Breathing exercises will be given 2 times a day, 5 repetitions, 2 sets. In addition to home-based conventional breathing exercises, coughing techniques and relaxation techniques will be taught and physical activity recommendations will be given.
  Interventions: Other: Conventional Breathing Exercises

INTERVENTIONS:
Other: Video Game-Based Breathing Exercises — The video game-based breathing exercises program will consist of 5 breathing games included in the BreathingLabs game kit and each game will be performed in 2 sets of 10 repetitions. The program will last for 8 weeks, 5 days a week, 30 minutes a day.
  Arms: Experimental Group
Other: Conventional Breathing Exercises — The conventional breathing exercises program will consist of routine breathing exercises. Breathing exercises will be given 2 times a day, 5 repetitions, 2 sets. The program will last for 8 weeks, 5 days a week, 30 minutes a day.
  Arms: Control Group

SUMMARY:
Conventional breathing exercises are recommended as a support to drug therapy, which is the primary treatment modality for symptom management in asthma patients. Video game-based applications are current approaches that enable exercises to be performed more fun, motivating, freely, and safely. The number of studies using video game-based approach as a respiratory exercise method is limited and no such study has been found in children with asthma. The aim of our study was to compare the effects of video game-based breathing exercises and conventional breathing exercises on pulmonary and extrapulmonary features in children with asthma.

Thirty-four children with asthma aged 8-18 years will be included in the study. Participants will be randomly divided into 2 groups as control group and experimental group. Demographic and clinical features of the patients will be recorded. Pulmonary function, respiratory muscle strength, dyspnea, fatigue, functional capacity, peripheral muscle strength, level of asthma control, and quality of life will be assessed by the spirometer, intraoral pressure measuring device, the Modified Borg Scale, the Fatigue Impact Scale, Spiropalm 6-min walk test, digital handheld manuel muscle tester, hydraulic hand dynamometer, asthma control test, and the Pediatric Quality of Life Inventory, respectively. Additionally, patient's adherence to the exercise program will be assessed by exercise diary. All assessments will be repeated before and after treatment.

Exercise training will be given to the patients for 8 weeks, 5 days a week, 30 minutes a day. The control group will receive home-based conventional breathing exercises; the experimental group will receive video game-based exercises consisting of breathing games. The exercise program will consist of the breathing games in the BreathingLabs game kit. In addition, relaxation techniques will be taught and physical activity recommendations will be given to the both groups.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years of age
* Being clinically diagnosed with asthma
* Being able to walk, cooperate, and clinically stable
* Having a computer, tablet, or mobile phone for the patients who will take part in the experimental group
* Volunteering to participate in the study

Exclusion Criteria:

* Upper respiratory tract infection or asthma attack in the last three weeks prior to participation in the study
* A history of hospitalisation within the last three weeks prior to participation in the study
* Having an upper respiratory tract infection or asthma attack or a history of hospitalisation during the exercise training programme
* Having a history of changes in medication used in the last three weeks prior to participation in the study
* History of previous lung or liver transplantation
* Having secondary diseases such as kyphoscoliosis etc. that may affect respiratory function
* Participation in ongoing or regular exercise training within the last 1 year
* Having completed less than 80% of the sessions that should be completed in total at the end of the treatment

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 8 weeks
  Forced Vital Capacity will be measured before six-minute walk test according to the guideline of (European Respiratory Society) ERS.
Forced Expiratory Volume in 1 second (FEV1) | 8 weeks
  Forced Expiratory Volume in 1 second will be measured before six-minute walk test according to the guideline of ERS.
Peak Expiratory Flow (PEF) | 8 weeks
  Peak Expiratory Flow will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Flow 25-75% (FEF25-75) | 8 weeks
  Forced Expiratory Flow 25-75% will be measured before six-minute walk test according to the guideline of ERS.
Maximal Inspiratory Pressure (MIP) | 8 weeks
  Maximal Inspiratory Pressure will be measured in accordance with American Thoracic Society (ATS)/ERS criteria using an electronic, mobile, (MicroRPM, Micro Medical; UK) intraoral pressure measuring device. Three measurements will be repeated for each maneuver and the highest value recorded as cmH2O.
Maximal Expiratory Pressure (MEP) | 8 weeks
  Maximal Expiratory Pressure will be measured in accordance with ATS/ERS criteria using an electronic, mobile, (MicroRPM, Micro Medical; UK) intraoral pressure measuring device. Three measurements will be repeated for each maneuver and the highest value recorded as cmH2O.
Level of Dyspnea | 8 weeks
  The dyspnea will be assessed by the Modified Borg Dyspnea Scale (MBS). The MBS is a 0 to 10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise or any activity. A score of 0 is given for no difficulty in breathing and a score of 10 is given for maximum difficulty in breathing.
Level of Fatigue | 8 weeks
  The fatigue will be assessed by the Fatigue Impact Scale (FIM). The FIM is a 40-item self-report questionnaire developed to measure the impact of fatigue on quality of life. There are 40 items, each of which is scored 0 (no problem) to 4 (extreme problem), providing a continuous scale of 0-160. It is composed of three subscales that describe how fatigue impacts upon cognitive (10 items), physical (10 items) and psychosocial functioning (10 items).
Spiropalm 6-minute Walk Test | 8 weeks
  To assess the functional capacity the 6-minute walk test (6MWT) will be performed. The 6MWT with Spiropalm 6 DYT (Cosmed, Spiropalm 6MWT) according to ATS guidelines. Walking distance, minute ventilation, respiratory rate, inspiratory capacity and breathing reserve will be recorded.
M. Quadriceps Muscle Strength | 8 weeks
  The m. quadriceps muscle strength will be measured using the MicroFet 2 hand-held dynamometer (Hogan Health Industries, USA). The test will be repeated three times for the dominant side and the average value in kilograms (kg) will be recorded.
M. Biceps Muscle Strength | 8 weeks
  The m. biceps muscle strength will be measured using the MicroFet 2 hand-held dynamometer (Hogan Health Industries, USA). The test will be repeated three times for the dominant side and the average value in kilograms (kg) will be recorded.
Handgrip Strength | 8 weeks
  The handgrip strength assessment will be performed with the Jamar hydraulic hand dynamometer (Performance Health; United States of America). The test will be repeated three times for both dominant and non-dominant hand and the average value in kilograms (kg) will be recorded.
Level of Asthma Control | 8 weeks
  The level of asthma control will be assessed by using the Asthma Control Test (ACT). The ACT is a patient self-administered tool for identifying those with poorly controlled asthma. The ACT assesses the frequency of shortness of breath and general asthma symptoms, use of rescue medications, the effect of asthma on daily functioning, and overall self-assessment of asthma control. The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Level of Quality of Life | 8 weeks
  The quality of life will be assessed by using the Pediatric Quality of Life Inventory (PedsQL). The PedsQL is a brief measure of health-related quality of life in children and adolescents and those with acute and chronic health conditions. Items on the PedsQL Scales are reverse scored and transformed to a 0-100 scale. Higher scores indicate better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hikmet Ucgun, PT, PhD, Principal Investigator — Atlas University
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No